CLINICAL TRIAL: NCT06123195
Title: Clinical, Biochemical, and Microbiological Effects of Constipation Treatment in Patients With Chronic Kidney Disease: A Pilot Feasibility Trial
Brief Title: Effects of Constipation Treatment in Chronic Kidney Disease: A Pilot Feasibility Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 23-09272-XP; R01DK135942 (NIH)
Record Dates: First submitted 2023-10-30; First posted 2023-11-08 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Chronic Kidney Disease; Constipation
Keywords: Chronic Kidney Disease; Constipation; Microbiota
MeSH Terms: conditions — Renal Insufficiency, Chronic; Constipation

STUDY DESIGN:
Intervention Model Description: A single-center, open-label, randomized, controlled, parallel-group, pilot feasibility trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Constipation treatment (Experimental): A 4-week intervention of constipation treatment with lactulose
  Interventions: Other: Constipation treatment
- Control (No Intervention): No constipation treatment except bisacodyl rescue therapy

INTERVENTIONS:
Other: Constipation treatment — Lactulose 15 mL (10 g) will be taken orally once daily (in the evening), which can be titrated at 1-week intervals in 15 mL (10 g) increments or decrements up to 60 mL (40 g) as a total daily dose.
  Arms: Constipation treatment

SUMMARY:
Constipation is one of the most prevalent gastrointestinal disorders in patients with chronic kidney disease (CKD) and has been associated with their adverse kidney and cardiovascular outcomes; however, little is known about the effects of constipation treatment on clinical outcomes nor on outcome-related biochemical and microbiological parameters in patients with CKD. The investigators aim to test the feasibility of delivering an intervention with constipation treatment and determine its effects on changes in clinical, biochemical, and microbiological parameters in patients with CKD and constipation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients >18 years old.
2. Patients able and willing to provide written informed consent and HIPAA authorization.
3. CKD stages G3-G5 without kidney replacement therapy with estimated glomerular filtration rate (eGFR) <60 mL/min/1.73m2 calculated using the Chronic Kidney Disease-Epidemiology Collaboration (CKD-EPI) 2021 creatinine equation.
4. Functional or opioid-induced constipation based on the Rome IV criteria.
5. Patients must refrain from taking any laxatives for at least one week prior to screening, although rescue with one bisacodyl 5 mg tablet will be allowed when a patient does not have a bowel movement for ≥3 consecutive days or when symptoms become intolerable.
6. A negative pregnancy test in female patients prior to enrolment, unless the patient is two years postmenopausal or has had a documented tubal ligation or hysterectomy.

Exclusion Criteria:

1. History of drug abuse, anorexia nervosa, or bulimia.
2. History of irritable bowel syndrome, inflammatory bowel disease, or Clostridium difficile bacterial infection (ever).
3. Liver cirrhosis or chronic active hepatitis (patients with treated hepatitis can be included).
4. Galactosemia.
5. Allergies to lactulose.
6. History of gastrointestinal surgery except appendectomy.
7. Use of antibiotics or immunosuppressants within 30 days prior to the enrollment in the study.
8. Use of pre- or probiotics within 30 days prior to enrollment in the study.
9. Women who are pregnant, capable of becoming pregnant and not participating in an acceptable form of birth control, or who are breast feeding.
10. Patients currently participating in another interventional study.
11. Major surgery within one month prior to enrollment in the study or planned surgery while the patient is in the study, other than dialysis vascular access surgery.
12. Patients who the investigator determine have a medical status that would preclude the patient's participation.
13. Patients on hemodialysis or peritoneal dialysis.
14. Patients with a functional kidney transplant.
15. Patients with past lactulose use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-11-17 (Actual); Study Completion 2025-11-17 (Actual)

PRIMARY OUTCOMES:
The feasibility of delivering the proposed interventions and performing the proposed examinations, assessed based on the adherence to prescribed protocol | From enrollment to the end of follow-up at 6 weeks
  The feasibility of delivering the applied interventions and performing the proposed examinations will be determined based on the following feasibility outcomes, assessed as 1) ≥90% of participants randomized in the intervention group and under observation will adhere to the proposed intervention, 2) ≥80% patients under observation will adhere to the study-specific timed collection of stool, urine, and blood samples, and 3) ≥85% patients will complete the study (<15% patients will be dropped out).

SECONDARY OUTCOMES:
Changes in serum creatinine | From enrollment to the end of follow-up at 6 weeks
  Changes in serum creatinine from baseline to 2, 4, and 6 weeks.
Changes in serum phosphorus | From enrollment to the end of follow-up at 6 weeks
  Changes in serum phosphorus from baseline to 2, 4, and 6 weeks.
Changes in serum p-cresyl sulfate and indoxyl sulfate | From enrollment to the end of follow-up at 6 weeks
  Changes in serum p-cresyl sulfate and indoxyl sulfate from baseline to 2, 4, and 6 weeks.
Changes in plasma potassium | From enrollment to the end of follow-up at 6 weeks
  Changes in plasma potassium from baseline to 2, 4, and 6 weeks.
Changes in plasma C-reactive protein | From enrollment to the end of follow-up at 6 weeks
  Changes in plasma C-reactive protein from baseline to 2, 4, and 6 weeks.
Changes in plasma lipopolysaccharide | From enrollment to the end of follow-up at 6 weeks
  Changes in plasma lipopolysaccharide from baseline to 2, 4, and 6 weeks.
Changes in urine albumin-creatinine ratio (UACR) and protein-creatinine ratio (UPCR) | From enrollment to the end of follow-up at 6 weeks
  Changes in urine albumin-creatinine ratio (UACR) and protein-creatinine ratio (UPCR) from baseline to 2, 4, and 6 weeks.
Changes in microbial parameters | From enrollment to the end of follow-up at 6 weeks
  Changes in gut and circulating microbiota from baseline to 2, 4, and 6 weeks.
Changes in stool consistency | From enrollment to the end of follow-up at 6 weeks
  Changes in stool consistency assessed by Bristol Stool Form Scale (BSFS) from baseline to 2, 4, and 6 weeks.
Changes in constipation symptoms | From enrollment to the end of follow-up at 6 weeks
  Changes in constipation symptoms assessed by Patient Assessment of Constipation Symptoms (PAC-SYM) score from baseline to 2, 4, and 6 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Memphis VA Medical Center, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No